CLINICAL TRIAL: NCT03623633
Title: Comparative Antiresorptive Efficacy of Alendronate or Raloxifene Following Discontinuation of Denosumab
Brief Title: Comparative Antiresorptive Efficacy Discontinuation of Denosumab
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joy Tsai, Assistant Professor, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018P001612
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Osteoporosis, Postmenopausal; Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Denosumab; Alendronate; Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Denosumab and Raloxifene (Active Comparator): denosumab and raloxifene
  Interventions: Drug: denosumab; Drug: raloxifene
- Denosumab and Alendronate (Active Comparator): denosumab and alendronate
  Interventions: Drug: denosumab; Drug: alendronate

INTERVENTIONS:
Drug: denosumab — denosumab 60 milligrams subcutaneously every 6 months
  Other Names: Prolia
Drug: alendronate — alendronate 70 milligrams weekly
  Other Names: Fosamax
  Arms: Denosumab and Alendronate
Drug: raloxifene — raloxifene 60 milligrams daily
  Other Names: Evista
  Arms: Denosumab and Raloxifene

SUMMARY:
Osteoporosis remains a significant healthcare burden for the United States. Current FDA-approved osteoporosis treatments include teriparatide, abaloparatide, bisphosphonates, denosumab, and raloxifene.

Denosumab is a fully human monoclonal antibody that specifically binds to receptor activator of nuclear factor kappa-B ligand (RANKL). Denosumab potently suppresses osteoclastic activity but bone turnover rapidly normalizes and bone turnover marker levels can rebound above baseline levels after the drug is discontinued.

This study will help us determine the optimal duration and relative efficacy of two oral antiresorptive medications that are FDA-approved for treatment of postmenopausal osteoporosis (alendronate and raloxifene) in preventing the rebound increase in bone turnover that occurs after denosumab discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* women aged 45+
* postmenopausal
* osteoporotic with high risk of fracture as per National Osteoporosis Foundation guidelines

Exclusion Criteria:

* no significant previous use of bone health modifying treatments
* hip fracture within one year of enrollment
* known congenital or acquired bone disease other than osteoporosis
* significant renal disease, liver disease, cardiopulmonary disease, or psychiatric disease
* abnormal calcium or parathyroid hormone level
* serum vitamin D <20 ng/dL
* anemia (hematocrit <32%)
* history of malignancy (except non-melanoma skin carcinoma)
* excessive alcohol use or substance abuse
* extensive dental work involving extraction or dental implant within the past 6 months or in the upcoming 12 months
* known contraindications to denosumab, alendronate, or raloxifene

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 51 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Serum c-telopeptide (CTX) | Month 12 to 18 months
  Change in serum CTX between month 12 and month 18
Bone mineral density (BMD) | Month 24 to 36 months
  Change in PA spine BMD between month 24 and month 36

CONTACTS AND LOCATIONS:
Overall Officials: Joy Tsai, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tsai JN, Jordan M, Lee H, Leder BZ. One versus 2 years of alendronate following denosumab: the CARD extension. Osteoporos Int. 2024 Dec;35(12):2225-2230. doi: 10.1007/s00198-024-07213-2. Epub 2024 Aug 7. PMID 39112628